CLINICAL TRIAL: NCT00378781
Title: Prospective, Randomized Trial Comparing Heparin and Minocycline-EDTA Flush for the Prevention of Catheter-Related Infections and Occlusions
Brief Title: Heparin or M-EDTA in Preventing Catheter-Related Infections and Blockages in Patients at High Risk for a Catheter-Related Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ID93-004; P30CA016672 (NIH); MDA-ID-93004 (Other: UT MD Anderson Cancer Center); CDR0000500199 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Cancer
Keywords: infection; poor vascular access; thromboembolism; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent breast cancer; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent small lymphocytic lymphoma; recurrent malignant testicular germ cell tumor; recurrent Wilms tumor and other childhood kidney tumors; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III ovarian epithelial cancer; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV ovarian epithelial cancer; stage IV small lymphocytic lymphoma; acute undifferentiated leukemia; mast cell leukemia; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; T-cell large granular lymphocyte leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; meningeal chronic myelogenous leukemia; prolymphocytic leukemia; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; adult grade III lymphomatoid granulomatosis; recurrent adult grade III lymphomatoid granulomatosis; childhood grade III lymphomatoid granulomatosis; recurrent childhood grade III lymphomatoid granulomatosis; Waldenstrom macroglobulinemia; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; primary central nervous system non-Hodgkin lymphoma; post-transplant lymphoproliferative disorder; intraocular lymphoma; stage I melanoma; stage II melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; metastatic childhood soft tissue sarcoma; nonmetastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; previously treated childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma; recurrent uterine sarcoma; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; localized osteosarcoma; metastatic osteosarcoma; recurrent osteosarcoma; chondrosarcoma; small intestine leiomyosarcoma; recurrent small intestine cancer; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Infections; Thromboembolism; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Breast Neoplasms; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Testicular Neoplasms; Wilms Tumor; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Biphenotypic, Acute; Leukemia, Mast-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Large Granular Lymphocytic; Leukemia, Prolymphocytic; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Waldenstrom Macroglobulinemia; Intraocular Lymphoma; Melanoma; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma; Chondrosarcoma | interventions — Heparin; Minocycline; Pentetic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Minocycline hydrochloride + Edetate Calcium Disodium (M-EDTA) flush solution into CVC once daily.
  Interventions: Drug: Minocycline-EDTA
- Arm II (Experimental): Heparin flush solution into CVC once daily.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin — Heparin flush solution into CVC once daily.
  Other Names: Hep-Lock
  Arms: Arm II
Drug: Minocycline-EDTA — M-EDTA flush solution into CVC once daily.
  Other Names: Minocycline hydrochloride; Edetate Calcium Disodium; M-EDTA
  Arms: Arm I

SUMMARY:
RATIONALE: Heparin or M-EDTA may prevent catheter-related infections and blockages in patients at high risk for a catheter-related infection. It is not yet known whether heparin is more effective than M-EDTA in preventing catheter-related infections and blockages in patients at high risk for a catheter-related infection.

PURPOSE: This randomized clinical trial is studying heparin to see how well it works compared with M-EDTA in preventing catheter-related infections and blockages in patients at high risk for a catheter-related infection.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the incidence of catheter-related infections (Staphylococcal and Candida) in patients at high risk for a catheter-related infection treated with heparin vs minocycline hydrochloride and edetate calcium disodium (M-EDTA).

Secondary

* Compare the incidence of catheter occlusions in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, prospective, multicenter study. Patients are stratified according to type of catheter (tunneled central venous catheter [CVC] vs nontunneled percutaneous CVC) and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive minocycline hydrochloride and edetate calcium disodium (M-EDTA) flush solution into the CVC once daily.
* Arm II: Patients receive heparin flush solution into the CVC once daily. Treatment in both arms continues for up to 3 months in the absence of unacceptable toxicity or until the removal of the catheter.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At high risk of acquiring a catheter infection, as evidenced by any of the following:

  * Diagnosis of leukemia, lymphoma, myeloma, or melanoma-sarcoma
  * Undergoing hematopoietic stem cell transplantation
  * Receiving aldesleukin
  * Pediatric cancer patients
* New (≤ 10 days old) functioning externalized tunneled or nontunneled central venous catheter (CVC), such as a Hickman/Broviac or Hohn catheter, or peripherally inserted central venous catheter (PICC) utilized for infusion of chemotherapy, blood and blood products, or other intermittent infusions

  * No occluded CVC
  * No existing local or systemic catheter infection

    * More than 3 days since removal of a prior CVC due to an infection
  * No externalized CVC that is projected to remain in place for < 2 weeks
  * No infusion ports or Groshong catheters
  * No coated CVC impregnated with an antimicrobial or antiseptic agent

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months
* No history of allergy to any tetracycline
* No contraindication to flush solution dwell time of ≥ 4 hours
* No hypocalcemia while receiving calcium supplementation through the catheter
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter-related infections during the study period (3 months) | 3 months

SECONDARY OUTCOMES:
Incidence of catheter occlusions during periods of prophylaxis (e.g., time period in which the catheter is locked with heparin or minocycline hydrochloride and edetate calcium disodium [M-EDTA]) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org